CLINICAL TRIAL: NCT06766630
Title: Exploring the Feasibility of Silk Fibroin Surgical Mesh in Rotator Cuff Tears Repair Enhancement
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Weiliang Shen, Ph.D., M.D. (Other)
Responsible Party: Sponsor-Investigator, Weiliang Shen, Ph.D., M.D., Director of Sports Medicine Department, the Second Affiliated Hospital of Zhejiang University School of Medicine, Second Affiliated Hospital, School of Medicine, Zhejiang University
Organization: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20241282
Record Dates: First submitted 2024-12-19; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- using silk fibroin surgical mesh to enhance rotator cuff tear repair (Experimental)
  Interventions: Device: Silk fibroin surgical mesh

INTERVENTIONS:
Device: Silk fibroin surgical mesh — This product is a mesh patch made of mulberry silk by warp knitting and degumming. The main component is fibroin protein

SUMMARY:
Rotator cuff tears result in shoulder joint pain and movement disorders, affecting patients' daily lives. The incidence rate rises with age and can be as high as 54% among people over 60 years old. Most rotator cuff tears are unable to heal spontaneously, and the tear area may gradually expand over time. Currently, the main surgical treatment for rotator cuff tears is to use suture anchors to stitch the rotator cuff tendon tissue back to the original anatomical insertion point. Large rotator cuff tears are often accompanied by fat infiltration and tendon retraction. When forcefully sutured, the tension is relatively high, which may lead to non-healing and re-tearing of the rotator cuff. Research indicates that the re-tear rate after rotator cuff tear repair is 20% - 30%, and this probability can reach 40% - 50% for large rotator cuff tears. For these irreparable and large tears, rotator cuff repair typically requires patch augmentation techniques. Surgeries are based on restoring the force couple effect of the rotator cuff as much as possible and covering it with repair materials to achieve reinforcement. Silk fibroin surgical mesh is made of silk fibroin which has good biocompatibility and can be generally placed in the area of rotator cuff tears that cannot be repaired through conventional surgeries. By providing support to the injured rotator cuff tissue, it improves the repair effect. It can reestablish the integrity of the rotator cuff, reducing mechanical tension at the repair site and maintaining the stability of the glenohumeral joint. Besides, it can also promote tissue healing, and cell infiltration and growth, thereby facilitating the biological repair of the injured rotator cuff and reducing the occurrence of postoperative re-tears.

ELIGIBILITY:
Inclusion Criteria:

* Preoperative:

  1. Age range of 50-75 years old (inclusive), gender not limited;
  2. Patients who require surgery due to rotator cuff tears detected by clinical and MRI examination;
  3. Evaluated as type IV and above according to Sugaya classification criteria;
  4. Patients with persistent or recurrent pain in the shoulder for more than 3 months;
  5. Full layer tendon tear of 1-5cm or full layer or complete tear of supraspinatus and/or infraspinatus tendon;
  6. History of non-surgical treatment failure;
  7. Understand the purpose of the trial, cooperate with surgical treatment and follow-up, voluntarily participate in the trial and sign an informed consent form;

     Intraoperative:
  8. Confirmed as a full-thickness tear of 1-5cm on the rotator cuff;
  9. Tendons can cover more than 50% of the humeral greater tuberosity of the shoulder joint.

Exclusion Criteria:

* 1. Pregnant and lactating women; 2.Individuals with contraindications for surgery or anesthesia, as well as those who are allergic to known ingredients of implanted products; 3. Unable to undergo MRI examination due to claustrophobia and other reasons; 4. Individuals with a history of rotator cuff repair on the affected side, or combined with other bone, joint, or muscle soft tissue injuries in the same limb; 5.Patients with subscapular muscle injury; 6.Those with any combination of diseases or symptoms that may affect the evaluation of efficacy, such as Hamada classification of grade 3 shoulder joint disease; 7.Those with residual rotator cuff tendon fatty infiltration ≥ grade 3 by Goutallier classification; 8.Individuals who have taken oral steroids or received steroid injections within 6 weeks prior to surgery; 9.Those who have participated in other interventional clinical trials within the past 3 months prior to the conduct of this trial; 10. Researchers believe that clinical trial participants who are not suitable for participation include but are not limited to those with uncontrolled blood sugar levels, heavy drinkers, smokers, and others who affect repair and healing.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2026-12-19 (Estimated)

PRIMARY OUTCOMES:
Re-tear rate at 12 months postoperatively | From enrollment to the end of treatment at 12 months

SECONDARY OUTCOMES:
Re-tear rate at 6 months postoperatively | From enrollment to 6 months after surgery
Constant-Murley Score postoperatively | From enrollment to the end of treatment at 12 months
Oxford Shoulder Score postoperatively | From enrollment to the end of treatment at 12 months
Degree of muscle atrophy | From enrollment to the end of treatment at 12 months
Fatty infiltration grading | From enrollment to the end of treatment at 12 months
Tendon thickness | From enrollment to the end of treatment at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided